CLINICAL TRIAL: NCT06256159
Title: Validity and Reliability of the 12-item Multiple Sclerosis Walking Scale (12-WS) in Subjects With Spinal Cord Injury
Acronym: 12-WS SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other); Swiss Paraplegic Research, Nottwil (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-02304
Record Dates: First submitted 2024-01-19; First posted 2024-02-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Spinal Cord Injuries; Gait Disorders, Neurologic
MeSH Terms: conditions — Spinal Cord Injuries; Gait Disorders, Neurologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with incomplete spinal cord injury (Other)
  Interventions: Other: 12 MSWS questionnaire

INTERVENTIONS:
Other: 12 MSWS questionnaire — The subject has to perform different gait assessments and fill out the 12-item multiple sclerosis walking scale questionnaire in one visit. Maximum 8 weekes after the first visit the subject has to fill out the same questionnaire again.

SUMMARY:
Established gait assessments for subjects with spinal cord injury (SCI) (6MWT, 10MWT, TUG, SCIM III and WISCI II) are widely used in the clinical and research setting. So far, no valid measurement exists that assesses the patients' perspective of walking ability in SCI. As there is the 12-item Multiple Sclerosis Walking Scale (12-WS) to assess the patients' perspective on gait ability in patients with multiple sclerosis, it is hypothesized that the 12-WS would also be a valid instrument for subjects with incomplete SCI. The main goal of this study is to collect data from clinical gait assessments in subjects with spinal lesions and to demonstrate that the 12-WS is a valid and reliable patient-reported outcome measurement for individuals with incomplete spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Diagnosis of chronic spinal cord injury (>6 months; cervical or thoracic motor incomplete traumatic or non-traumatic (AIS C, D) above T12
* Must have impaired walking function as demonstrated by neurological examination.

Exclusion Criteria:

* Women who are pregnant or breast feeding
* Current orthopaedic problems of lower limbs
* History of major cardiac condition (e.g., infarction, insufficiency (NYHA II-IV))
* History of major pulmonary condition (e.g., chronic obstructive pulmonary disease GOLD II-IV
* Current major depression or psychosis
* Participation in another interventional study (except specTra-study) that may have an impact on walking function.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Re-test reliability of the subjective perceived limitations in ambulation of the 12-item Multiple Sclerosis Walking Scale (12-WS) in subjects with incomplete SCI. | Change from day 1 to day 2
  The scale is numeric and ranges from 0-100. A lower score means a better outcome.
Validity of the 12-item Multiple Sclerosis Walking Scale (12-WS) in subjects with incomplete SCI. | Day 1
  The scale is numeric and ranges from 0-100. A lower score means a better outcome.

SECONDARY OUTCOMES:
Clinical examination (a neurological examination including the ASIA score (categoric outcome grade A-E) - International Standards for Neurological Classification of Spinal Cord Injury | Day 1
  Grade "A" means most impaired, grade "E" means less impaired.
Walking impairment (numeric value from 0-20) - WISCI II | Day 1
  The scale is numeric and ranges from 0-20. A higher score means a better outcome.
Walking distance (m) and number of rests - 6MWT | Day 1
  High distance and low number of rests means better outcome.
Walking speed (m/s) - 10-meter walkint test (10MWT) | Day 1
  High speed means better outcome.
Walking speed including sit-stand transfer (s) - Timed Up and Go-test (TUG) | Day 1
  The fewer seconds needed, the better the outcome.
Functional independence (numeric value from 0-40) - Spinal Cord Independence Measure III (SCIM III), Items 9-17 | Day 1
  The scale is numeric and ranges from 0-30). A higher score means a better outcome.
Dynamic balance (numeric value from 0-30) - Functional Gait Assessment (FGA) | Day 1
  The scale is numeric and ranges from 0-30). A higher score means a better outcome.
Change in impairment level (nominal outcome Yes - No) - Follow up questions in telephone interview | Day 2, maximum 8 weeks after day 1
  Only subjects with NO changes in impairment level will be used for reliability testing.

CONTACTS AND LOCATIONS:
Overall Officials: Björn Zörner, PD Dr., Principal Investigator — University of Zurich
Locations (2):
- Switzerland (2):
  - Swiss Paraplegic Center, Nottwil
  - Balgrist University Hospital, Zurich